CLINICAL TRIAL: NCT05779345
Title: Clinical and Radiographic Evaluation of Stability of Short Implants Versus Standard Blx Implants Placed With Internal Sinus Floor Elevation in Posterior Maxilla: A Randomized Controlled Clinical Trial
Brief Title: Stability of Short Implants Versus Standard Blx Implants With Internal Sinus Floor Elevation in Posterior Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hani Elnahass, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short implants (Active Comparator): short 6 mm straumann blx implants
  Interventions: Procedure: surgery
- regular length + internal sinus lift (Active Comparator): regular length implant 10 mm, in addition to internal sinus lift procedure
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — short implant placement

SUMMARY:
Implants in the maxillary posterior region are associated with compromised bone in both quantity - notably in vertical dimension- and quality. Along with the fact that the posterior teeth are subjected to higher occlusal forces than the anterior teeth (Marianne Morand & Tassos Irinakis, 2007). In order to overcome these shortcomings, various procedures have been advocated including open and closed sinus lift (Nkenke E & Stelzle F, 2009; Schropp et al, 2003). The use of short implants is a valid alternative for these procedures (Wallace SS & Froum SJ, 2003) sparing the need of applying augmentation techniques with the associated increased time, morbidity and complexity of such procedures.

DETAILED DESCRIPTION:
To overcome anatomical and physiological limitations, different sinus augmentation techniques with immediate or delayed (6-8 months post augmentation) implant placement have been proposed. The most common one is the sinus elevation with a lateral window approach. Although these protocols evoke a high level of success in augmenting the bone quantity (Nkenke E & Stelzle F, 2009; Schropp et al, 2003) many patients refuse them because of the invasiveness of the augmentative procedure, with obvious prolonged healing times and increased morbidity and costs (Fugazzotto, 2003; Bra¨gger et al, 2004; Toffler, 2004). An alternative therapy for restoring areas of limited bone dimension is the placement of short implants (Wallace SS & Froum SJ, 2003). ''Standard length implants'' are those of 10 mm in length and have been defined as the minimal length for anticipated success (Griffin TJ & Cheung WS, 2004).

ELIGIBILITY:
Inclusion Criteria:

* Single edentuolous site at maxillary posterior region
* The available bone height below the maxillary sinus should be 7-8mm
* Patients ≥ 20 years old
* Bucco-palatal bone width should be ≥6mm
* Adequate interarch space
* Bounded, single

Exclusion Criteria:

* Patients with local pathological defects related to the area of interest.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as alcoholism or parafunctional habits.
* Inadequate inter-arch space for implant prosthetic part
* Smokers
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-04-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
crestal bone level | 1 year
  crestal bone level will be assessed by periapical standardized radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Hani El Nahass, Professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Greater Cairo, Egypt